CLINICAL TRIAL: NCT04732130
Title: Longitudinal Monitoring During Different Intermittent Fasting Protocols in Non-Obese Adults - A Randomized Clinical Trial
Brief Title: Monitoring During Different Intermittent Fasting Protocols in Non-Obese Adults
Acronym: LIMITFOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipp Gerber (Other)
Responsible Party: Sponsor-Investigator, Philipp Gerber, MD, MSc, Senior Physician / Group Leader, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIMITFOOD
Record Dates: First submitted 2021-01-19; First posted 2021-02-01 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Intermittent Fasting; Overweight; Time Restricted Feeding
MeSH Terms: conditions — Intermittent Fasting; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time-Restricted Feeding (Active Comparator): Participants in the time-restricted feeding are instructed to eat ad libitum from 12:00 to 20:00 daily, and fast from 20:00 to 12:00 daily for 4 weeks.
  Interventions: Behavioral: Time-Restricted Feeding
- Alternate Day Fasting (Active Comparator): Participants in the alternate day fasting group are instructed to eat every second day ad libitum, but to abstain from calorie intake on fast days (100 % restriction) for 4 weeks.
  Interventions: Behavioral: Alternate Day Fasting
- Control (No Intervention): Participants in the control group are instructed to maintain their habitual diet regimen.

INTERVENTIONS:
Behavioral: Time-Restricted Feeding — Participants are instructed to limit food intake to maximum 8 hours per day.
  Arms: Time-Restricted Feeding
Behavioral: Alternate Day Fasting — Participants are instructed to fast every other day.
  Arms: Alternate Day Fasting

SUMMARY:
LIMITFOOD is a randomized clinical intervention study that investigates the effects of two different intermittent fasting protocols compared to a control group on the health of normal- and overweight adults. A total of 72 participants will be randomized into three equally sized groups: an alternate day fasting, a time-restricted feeding and a control group.

DETAILED DESCRIPTION:
The prevalence of overweight has risen considerably all over the world in the past century. Epidemiological studies have shown that, starting from a body mass index of 20-21 kg/m2, increasing BMI levels are associated with progressively increased risks of developing diabetes, cardiovascular disease, several types of cancer and other diseases. The problem is pronounced by the unlimited and constant availability of food. Treatment of overweight is still difficult and finding effective and more personalized strategies to manage these conditions is crucial.

Intermittent fasting has been suggested as an alternative way to address these problems. Intermittent fasting is an eating pattern that involves rotating periods of eating and fasting. Animal studies and previous human clinical trials have provided evidence that various types of intermittent fasting lead to weight loss and improved health markers not only in obese, but also in healthy, non-obese adults.There are several types of intermittent fasting. The most popular version is time-restricted feeding (TRF), which allows ad libitum (at one's pleasure) energy intake within a defined period of time each day (6-12h). Another subtype of IF is called alternate day fasting (ADF). ADF is defined as 'feast days' on which food is consumed ad libitum, which alternate with 'fast days' on which food is withheld or reduced.

However, despite the growing popularity of intermittent fasting, it is not clear which type of IF is most effective and what fasting window is needed to induce beneficial effects. Additionally, tools to longitudinally track personal progress of dieting are lacking. Therefore, the main objective of this study is to compare the effects of each of two different intermittent fasting protocols (TRF and ADF) on metabolic parameters to a control group. Furthermore, a new dynamic measurement technique, using breath analysis, will allow to better monitor the progress of individual participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years, both inclusive
* Non-obese, BMI between 23 and 30 kg/m2, both inclusive
* Non-smoker
* Good knowledge of German or English language
* Stable weight change (change < +/- 10% current bodyweight) for 3 months prior to the study
* Glycohemoglobin (HbA1c) < 5.7% without glucose lowering medication
* LDL-cholesterol < 180 mg/dl without lipid lowering medication
* Blood pressure < 140/90 mmHG without blood pressure lowering medication

Exclusion Criteria:

* Subjects who have a fasting period of > 12h per day on a regular basis and do not eat at least three main meals per day.
* Current habitual use of dietary supplements (e.g. vitamins, minerals) and/or unwillingness to cease intake of dietary supplements.
* Antibiotics intake during 3 months prior to the study
* Food intolerances, allergies and sensitivities (e.g. lactose/gluten intolerance, food allergies) or dietary restrictions (e.g. vegan lifestyle)
* Acute or chronic infections, malignant disease, renal, hepatic (more than two-fold increased transaminases), pulmonary, neurological (epilepsy) or psychiatric diseases, manifested atherosclerosis, or any other disease precluding participation in the study.
* Diabetes
* Known alcohol, substance or drug abuse, concomitant medication
* More than four hours of physical exercise per week
* Women who are pregnant, breast-feeding or aiming to become pregnant during course of the trial
* Women and men on hormonal supplementation
* Women with a very irregular menstrual cycle
* Therapy with antidepressants within the past 6 months
* Regular therapy with acetylsalicyclic acid or current medication to regulate blood sugar, blood pressure or lipids
* Subjects likely to fail to comply with the study protocol
* Subjects who do not give informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Fat mass | 4 weeks
  Change in whole body fat mass

SECONDARY OUTCOMES:
Continuous glucose monitoring (CGM) | 4 weeks
  During the study period the CGM system will measure the continuous glucose concentration of the participants and thereby any changes will be measured.
Physical activity energy expenditure | 4 weeks
  Change in mean physical activity energy expenditure will be recorded using an Actiheart monitor during the intervention.
Resting metabolic rate (measured by indirect calorimetry) | 4 weeks
  Change in resting metabolic rate

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Gerber, MD, Principal Investigator — University of Zurich
Locations (1):
- Department of Endocrinology, Diabetology and Clinical Nutrition, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derron N, Guntner AT, Weber IC, Braun J, Koska IO, Othman A, Monch L, von Eckardstein A, Puhan MA, Beuschlein F, Hochuli M, Zamboni N, Guggenberger R, Gerber PA. Alternate-day fasting elicits larger changes in fat mass than time-restricted eating in adults without obesity - A randomized clinical trial. Clin Nutr. 2025 Oct;53:212-221. doi: 10.1016/j.clnu.2025.08.033. Epub 2025 Sep 3. PMID 40945487